CLINICAL TRIAL: NCT02967887
Title: Single-arm, Prospective, Multicenter Clinical Trial to Assess the Efficacy and the Safety of Combination Therapy of Hepatic Arterial Infusion of Cisplatin and 5-FU in Advanced Hepatocellular Carcinoma With Low Expression of HMGB2 Biomarker
Brief Title: Evaluation of Hepatic Arterial Infusion of Cisplatin and 5-FU in Biomarker Stratified HCC
Acronym: SHINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CbsBioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBS-PCT-01
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Carcinoma Non-Resectable
MeSH Terms: interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cisplatin and 5-fluorouracil (Experimental): Enrolled patients with pre-treatment tumor biopsy will receive Cisplatin (60mg/m2 for 2h on day 2) and 5-fluorouracil (500mg/m2 for 5h on days 1-3) through implanted port system. This treatment will be repeated every 4 weeks, up to 6 times.
  Interventions: Drug: cisplatin and 5-fluorouracil

INTERVENTIONS:
Drug: cisplatin and 5-fluorouracil — Hepatic arterial infusion of Cisplatin (60mg/m2 for 2h on day 2) and 5-fluorouracil (500mg/m2 for 5h on days 1-3) through implanted port system (chemoport)
  Other Names: CBD-01 and CBD-02

SUMMARY:
This study is to assess the efficacy and the safety of hepatic arterial infusion of cisplatin and 5-fluorouracil (HAIC) in advanced HCC patients stratified by biomarker expression predicting therapeutic response.

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) with cisplatin and 5-fluorouracil has been used in advanced HCC. However, cisplatin or 5-fluorouracil acts on cells without tumor selectivity. Therefore, to improve the tumor selectivity and effectiveness of HAIC, molecular subtyping-based stratification strategies should be considered. In this study, patients who have progressed or intolerance to sorafenib with non-metastatic HCC in TNM stage III-IVA and ECOG PS 0 or 1, Child-Pugh class A will be enrolled. 96 patients with pre-treatment tumor biopsy will receive Cisplatin (60mg/m2 for 2h on day 2) and 5-fluorouracil (500mg/m2 for 5h on days 1-3) through implanted port system. This treatment will be repeated every 4 weeks, up to 6 times. The primary objective is to determine overall response rate, where benefit is defined as complete or partial response according to mRECIST V1.1. Secondary endpoints include time to progression, progression free survival. The biopsy tissue will be subjected to real time reverse transcriptase polymerase chain reaction for quantification of gene expression levels. Patients will be categorized into two groups according to gene expression results, and then AUC value of ROC curve analysis will be evaluated as an exploratory endpoint to assess predictive performance of biomarker for therapeutic response of HAIC.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* Patients with advanced hepatocellular carcinoma who have progressed or intolerance to Sorafenib
* Patients with advanced hepatocellular carcinoma who cannot be treated with surgery, transplantation, RFA, or TACE.
* TNM stage III/IV (including intrahepatic single or multiple tumors without extrahepatic metastasis regardless of lymph node metastasis)
* ECOG performance status of 0 or 1
* Liver function status of Child-Pugh Class A or B
* more than 3 months of life expectancy
* serum creatinine <1.5 mg/dL
* aminotransferase <5 times the upper limit of normal
* absolute neutrophil count >1,500 cells/lL
* platelet count >75,000/lL
* hemoglobin >10 g/dL

Exclusion Criteria:

* patients with extrahepatic tumors
* Patients requiring combined treatment with chemotherapy, radiotherapy, TACE, RFA, or others
* Patients in any severe and/or uncontrolled medical conditions
* patients with history of allergic response to CT contrast media
* patients who participated as subjects in other interventional clinical studies (as of the date of visit) within 60 days before drug administration
* Any person deemed inappropriate by reason of the investigator for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response | Approximately 6 months
  Objective tumor response according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST) assessed by radiological review

SECONDARY OUTCOMES:
Time-to-Progression | Approximately 24 months
Progression-free-survival | Approximately 24 months

OTHER OUTCOMES:
Exploratory endpoint: Diagnostic performance of biomarkers | Through study completion, an average of 3 months
  Patients will be categorized according to the result of biomarker expression and then AUC value of ROC curve analysis will be evaluated as an exploratory endpoint to assess predictive performance of biomarkers for therapeutic response of drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Si Hyun Bae, MD., PhD., Principal Investigator — The Catholic University of Korea
Locations (12):
- South Korea (12):
  - Korea University Ansan Hospital, Ansan
  - Sooncheonhyang University Hospital Bucheon, Bucheon-si
  - The Catholic University of Korea Bucheon ST. Mary's Hospital, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Sooncheonhyang University Hospital Seoul, Seoul
  - The Catholic University of korea, Seoul ST. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea ST. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided